CLINICAL TRIAL: NCT03748394
Title: Enhancing Work Ability in Common Mental Disorders: Comparing Two Interventions in Primary Care Rehabilitation
Brief Title: Interventions to Facilitate Working While Depressed and Anxious
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGFOUREG-588531
Record Dates: First submitted 2016-12-28; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Work Capacity
Keywords: Work capacity evaluation; Common mental disorders; Occupational therapy; Physical Therapy Modalities
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Work-directed rehabilitation (Experimental): Work-directed, person-centered plan using modules of occupational therapy and physical therapy
  Interventions: Behavioral: Work-directed rehabilitation
- Physical activity (Active Comparator): Physical activity according to national health recommendations
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Work-directed rehabilitation — Each participant starts with a meeting together with an occupational therapist or a physical therapist, focusing on the participant's resources and obstacles for functioning well at work. A plan is designed and carried out over 8 weeks, including 1-4 different treatment modules of occupational and physical therapy, to support the person's ability to function at work
  Arms: Work-directed rehabilitation
Behavioral: Physical activity — In a meeting with a physical therapist, each participant receives advice on physical activity to support mental health, according to national recommendations. The participant is offered to train at a local gym during 8 weeks.
  Arms: Physical activity

SUMMARY:
The study compares the effects of two add-on interventions in primary care rehabilitation, on work ability and psychological health, in workers with common mental disorders. One intervention consists of a person-centered plan using work-directed treatment modules of occupational therapy and physical therapy, during 8 weeks. The other intervention consists of supported physical activity during 8 weeks. The primary outcome is work ability, measured by the work ability index and days on sick leave.

DETAILED DESCRIPTION:
Common mental disorders (CMD), including mild to moderate depression, anxiety disorders and exhaustion disorder, are a major cause of sick leave and work disability. Compared to other disorders, work-related problems associated with CMD is sparsely explored. While recommended treatments, such as antidepressants or cognitive behavioral therapy have effects on psychiatric symptoms, the effect on work capacity is unclear, suggesting a need for alternative interventions.

The aim of this study is to evaluate the effects of an add-on work-directed intervention in primary care rehabilitation, compared to a physical activity control, for persons with CMD.

The goal of the experimental condition is to enhance the participant's ability to work by creating an individually tailored plan for self-management, supported by occupational and physical therapy techniques, such as structuring daily activities, stress management or body awareness techniques. Enhancing self-management is the core of this intervention and also a new approach compared to earlier efforts to promote work capacity.

ELIGIBILITY:
Inclusion Criteria:

* Unipolar depression or anxiety disorder according to the Mini Neuropsychiatric Interview (DSM-5 criteria).
* Currently working to some extent, part time sick leave is accepted.

Exclusion Criteria:

* Substance abuse according to the Mini interview
* High suicide risk according to the Mini interview
* Psychotic symptoms according to the Mini interview

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Work ability | change in score from baseline to 8 weeks
  Work Ability Index

SECONDARY OUTCOMES:
Depression severity | change in score from baseline to 8 weeks
  Montgomery Asberg Depression Rating Scale
Anxiety symptoms | change in score from baseline to 8 weeks
  Beck Anxiety Index
Mental wellbeing | change in score from baseline to 8 weeks
  WHO-5 Mental Wellbeing Index

CONTACTS AND LOCATIONS:
Overall Officials: Gunnel Hensing, Professor, Principal Investigator — Göteborg University
Locations (1):
- Närhälsan Gibraltar Rehabmottagning, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No